CLINICAL TRIAL: NCT00487032
Title: A Proof of Concept Study to Evaluate Differential Tachyphylaxis of Alpha 1 and Alpha 2 Adrenoreceptor Mediated Decongestant Response to Oxymetazoline and Its Acute Reversal by Corticosteroid in Healthy Volunteers
Brief Title: Differential Adrenoreceptor Mediated Tachyphylaxis and Upregulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brian J Lipworth (Other)
Responsible Party: Sponsor-Investigator, Brian J Lipworth, Professor (Clinical) Airway allergy and COPD, University of Dundee
Organization: University of Dundee (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: VAI03; 2007-003194-82
Record Dates: First submitted 2007-06-14; First posted 2007-06-15 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Allergic Rhinitis; Tachyphylaxis; Rhinitis Medicamentosa
Keywords: allergic rhinitis; rhinitis medicamentosa; imidazolines; corticosteroid
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Oxymetazoline; Prazosin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Prazosin 1mg challenge to block alpha 1 adrenoreceptors
  Interventions: Drug: Oxymetazoline 0.05% w/v; Drug: Fluticasone propionate 50 micrograms per actuation; Drug: Prazosin hydrochloride
- 2 (Placebo Comparator): Placebo to Prazosin
  Interventions: Drug: Placebo to Prazosin

INTERVENTIONS:
Drug: Oxymetazoline 0.05% w/v — 2 squirts in each nostril thrice daily
  Arms: 1
Drug: Fluticasone propionate 50 micrograms per actuation — 2 Squirts in each nostril twice daily
  Arms: 1
Drug: Prazosin hydrochloride — Prazosin 1mg one dose only
  Arms: 1
Drug: Placebo to Prazosin — Placebo 1 tablet one dose only
  Arms: 2

SUMMARY:
The investigators wish to evaluate the onset of tolerance to nasal decongestants like oxymetazoline (available over the counter) and the mechanism of tolerance particularly with differential effects on alpha 1 and alpha 2 adrenoreceptors on the nose. The investigators will 'tease' out by using an alpha 1 blocker called Prazosin. The investigators hypothesize that alpha 1 receptors mediate arterial constriction and this will be captured by measuring nasal blood flow. The investigators also hypothesize that alpha 2 receptors mediate venous sinusoid constriction and this the investigators will capture by airflow parameters like Peak Nasal Inspiratory Flow, Rhinomanometry, Oscillometric indices etc.

DETAILED DESCRIPTION:
Allergic rhinitis affects upto 25% of the worldwide population and is associated with asthma. Furthermore, nonallergic rhinitis accounts for more than 50% of Rhinitis sufferers. Patients with Allergic Rhinitis, Nonallergic Rhinitis and Common cold have nasal blockage as their principal symptom. Nasal blockage can affect sleep quality and impairs daytime performance. It is a major cause of sickness absenteeism and has been shown to adversely affect quality of life. The most efficacious class of drugs for this symptom are the nasal decongestants (sympathomimetics acting on alpha receptors). Unfortunately prolonged use of these sprays can result in a condition of tolerance (reduced efficacy), rebound nasal congestion and nasal hyperreactivity called Rhinitis Medicamentosa. It is a poorly understood condition and the mechanism of action is unclear. What is also not clear is the time to onset of tolerance. Finally many research studies have demonstrated that use of these nasal sprays for many weeks did not result in any side effects. Although evidence for this is conflicting, in vitro studies have shown that adrenoreceptors are known to develop tolerance within days of agonist use. Moreover beta adrenoreceptors in the lung can be upregulated (i.e., tolerance can be reversed) by use of corticosteroids. We have also seen over many years of clinical practise that concomitant use of steroid sprays and decongestants does not result in tolerance or rebound. Finally, research has shown that rebound congestion can be treated by stopping the decongestant spray and starting steroid sprays. We are not studying rebound congestion which takes years of decongestant abuse to develop. What we would like to demonstrate is the onset of tolerance (which precedes rebound) and its reversal by steroids. We would also find out if one of the two alpha receptors is responsible for this, which may lead to a selective alpha 1 or alpha 2 agonist being used safely in the nose.We, therefore propose to conduct a proof of concept study to evaluate the onset of tolerance by nasal decongestant Oxymetazoline (OXY, its differential effects on alpha 1 and alpha 2 adrenoreceptors by an alpha 1 blocker Prazosin and finally the reversal of this process by intranasal steroid (Fluticasone). We are recruiting 31 patients (38 to complete 31) according to previous research studies and PNIF as an outcome measure if the true difference between the two arms is 10L/min. There would be a total of 7 visits to the Asthma and Allergy group at Ninewells Hospital, Dundee and Perth Royal Infirmary. Healthy Volunteers from 18-65 years of age will attend for a screening visit. Their Peak Nasal Inspiratory Flow (PNIF) must be more than 100L/min (best of three). All patients who satisfy the inclusion criteria and none of the exclusion criteria will be included in the trial. They will be issued a Peak Nasal Inspiratory Flow diary and a symptom diary. This they will record at home each morning before and 20 min after using their nasal sprays and repeated before bedtime. They will be issued with Oxymetazoline nasal spray to be used according to the recommended dose of 2 squirts in each nostril three times daily (can be used upto four times daily), on waking up, after lunch and before bedtime. The first visit will include a baseline nasal blood flow and airflow tests. The order of the tests will be as follows: Firstly, nasal peak inspiratory flow (PNIF), secondly, active anterior rhinomanometry, thirdly, nasal impulse oscillometry, and finally, nasal blood flow using Laser Doppler Flowmetry. They will also have lying/standing blood pressure measurements. This will be followed by the administration of 1mg of oral Prazosin/Placebo in a supine position. 3 hours later a dose response curve (DRC) will be constructed with OXY at 20 minute intervals using cumulative sequential doses of 50 µg [1 squirt] , 100 µg[+ 1 squirt ] and 200 µg per nostril[+ 2 squirts].After 1st dose and 2nd dose, only PNIF and Rhinomanometry will be performed 10 minutes after each dose administration . After the last dose, the order of tests will be again PNIF, active anterior rhinomanometry, nasal impulse oscillometry, and laser Doppler flowmetry. For the first 2 hours lying/standing BP will be measured at ½ hourly intervals; hourly thereafter. They will be asked to lie down till the end of the visit (4 hours down) or until no postural drop in blood pressure is recorded whichever comes first. There is very rarely a drop in blood pressure on giving Prazosin called 'First Dose Hypotension'. This happens in hypertensive patients who take a high dose of an alpha blocker like Prazosin. Therefore the British National Formulary will advise patients to be given a dose of say 0.5 milligrammes thrice daily with the first dose at bedtime and them slowly increased to upto a maximum daily dose of 20 milligrammes. We are within this dose range. Moreover, in clinical practise, doses of upto 5 milligrammes have been prescribed and in previous research trials upto 10 milligrammes have been given to Healthy Volunteers who have a lesser risk of this first dose effect. Moreover, according to previous pharmacokinetic and pharmacodynamic studies within 4-6 hours Prazosin effect on Blood Pressure wanes. Therefore we would conduct the Prazosin challenge test and the OXY dose response in a supine position and no patient will be discharged till the postural BP change is within normal limits. Laser Doppler Flowmetry is a noninvasive test designed to measure blood flow through the nose. Rhinomanometry is another noninvasive test measuring nasal resistance and flow. Oscillometry is another parameter measured on the Rhinomanometry machine itself.PNIF is a noninvasive measure of airflow which is basically a peak flow meter reversed. Thus no invasive measures will be used. This order of tests will be performed on Day 1 and repeated on Day 14 to compare acute with chronic agonist use. On day 14 Fluticasone nasal spray 2 squirts twice daily will be issued and on Day 17 the same order of tests will be performed. As this is a cross over study the patients receiving placebo will have prazosin in the second arm following a weeks washout in between. The same procedure for Prazosin/Placebo challenge will be followed throughout.

ELIGIBILITY:
Inclusion Criteria:

* Male of Female aged 18-65 years.
* Healthy volunteers with a negative history of seasonal or perennial nasal symptoms other than occasional common colds. Atopy will not preclude inclusion into the study as long as patients have no nasal symptoms.
* Current non-smokers (ex-smokers for greater than 6 months duration with a total smoking history of less than 5 pack-years will be eligible).
* PNIF > 100L/min (best effort of 3) and reversibility with OXY 2 squirts in each nostril (20 min reading) > 20 L/min.
* Ability to give a written informed consent.
* Ability and willingness to comply with the requirements of the protocol.

Exclusion Criteria:

* Recent respiratory tract/sinus infection within the last 2 months.
* Pregnancy, planned pregnancy or lactation.
* Known or suspected hypersensitivity to any of the IMP's.
* Concomitant use of medicines (prescribed, OTC or herbal) like alpha blockers that may interfere with the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the difference in peak PNIF response to incremental doses of Oxymetazoline [i.e. as a dose response] | 1 hour

SECONDARY OUTCOMES:
Active Anterior Rhinomanometry | 1 hour
Nasal oscillometric indices | 1 hour
Laser Doppler Flowmetry to measure nasal blood flow | 1 hour
Systolic, Diastolic blood pressure(measure of alpha blockade) | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Vaidyanathan, MRCS, DOHNS, Principal Investigator — University of Dundee; Brian Lipworth, MD, FRCP, Study Director — University of Dundee
Locations (2):
- United Kingdom (2):
  - Perth Royal Infirmary (Tayside NHS Trust), Perth, Perthshire
  - Ninewells Hospital and Medical School (Tayside NHS Trust, University of Dundee), Dundee, Tayside

REFERENCES:
- [Background] Bousquet J, Van Cauwenberge P, Khaltaev N; Aria Workshop Group; World Health Organization. Allergic rhinitis and its impact on asthma. J Allergy Clin Immunol. 2001 Nov;108(5 Suppl):S147-334. doi: 10.1067/mai.2001.118891. No abstract available. PMID 11707753
- [Background] Nassef M, Shapiro G, Casale TB; Respiratory and Allergic Disease Foundation. Identifying and managing rhinitis and its subtypes: allergic and nonallergic components--a consensus report and materials from the Respiratory and Allergic Disease Foundation. Curr Med Res Opin. 2006 Dec;22(12):2541-8. doi: 10.1185/030079906x158057. PMID 17265594
- [Background] Nolte H, Nepper-Christensen S, Backer V. Unawareness and undertreatment of asthma and allergic rhinitis in a general population. Respir Med. 2006 Feb;100(2):354-62. doi: 10.1016/j.rmed.2005.05.012. Epub 2005 Jul 11. PMID 16005621
- [Background] Gupta R, Sheikh A, Strachan DP, Anderson HR. Burden of allergic disease in the UK: secondary analyses of national databases. Clin Exp Allergy. 2004 Apr;34(4):520-6. doi: 10.1111/j.1365-2222.2004.1935.x. PMID 15080802
- [Background] Ferguson BJ. Influences of allergic rhinitis on sleep. Otolaryngol Head Neck Surg. 2004 May;130(5):617-29. doi: 10.1016/j.otohns.2004.02.001. PMID 15138430
- [Background] Patou J, De Smedt H, van Cauwenberge P, Bachert C. Pathophysiology of nasal obstruction and meta-analysis of early and late effects of levocetirizine. Clin Exp Allergy. 2006 Aug;36(8):972-81. doi: 10.1111/j.1365-2222.2006.02544.x. PMID 16911353
- [Background] Hadley JA. Cost-effective pharmacotherapy for inhalant allergic rhinitis. Otolaryngol Clin North Am. 2003 Oct;36(5):825-36. doi: 10.1016/s0030-6665(03)00054-9. PMID 14743775
- [Background] Graf P. Long-term use of oxy- and xylometazoline nasal sprays induces rebound swelling, tolerance, and nasal hyperreactivity. Rhinology. 1996 Mar;34(1):9-13. PMID 8739860
- [Background] Scadding GK. Rhinitis medicamentosa. Clin Exp Allergy. 1995 May;25(5):391-4. doi: 10.1111/j.1365-2222.1995.tb01068.x. No abstract available. PMID 7553240
- [Background] Ramey JT, Bailen E, Lockey RF. Rhinitis medicamentosa. J Investig Allergol Clin Immunol. 2006;16(3):148-55. PMID 16784007
- [Background] Petruson B. Treatment with xylometazoline (Otrivin) nosedrops over a six-week period. Rhinology. 1981 Sep;19(3):167-72. PMID 6171024
- [Background] Yoo JK, Seikaly H, Calhoun KH. Extended use of topical nasal decongestants. Laryngoscope. 1997 Jan;107(1):40-3. doi: 10.1097/00005537-199701000-00010. PMID 9001263
- [Background] Watanabe H, Foo TH, Djazaeri B, Duncombe P, Mackay IS, Durham SR. Oxymetazoline nasal spray three times daily for four weeks in normal subjects is not associated with rebound congestion or tachyphylaxis. Rhinology. 2003 Sep;41(3):167-74. PMID 14579657
- [Background] Andersson KE, Bende M. Adrenoceptors in the control of human nasal mucosal blood flow. Ann Otol Rhinol Laryngol. 1984 Mar-Apr;93(2 Pt 1):179-82. doi: 10.1177/000348948409300216. PMID 6201119
- [Background] Corboz MR, Rivelli MA, Varty L, Mutter J, Cartwright M, Rizzo CA, Eckel SP, Anthes JC, Hey JA. Pharmacological characterization of postjunctional alpha-adrenoceptors in human nasal mucosa. Am J Rhinol. 2005 Sep-Oct;19(5):495-502. PMID 16270605
- [Background] Michelotti GA, Price DT, Schwinn DA. Alpha 1-adrenergic receptor regulation: basic science and clinical implications. Pharmacol Ther. 2000 Dec;88(3):281-309. doi: 10.1016/s0163-7258(00)00092-9. PMID 11337028
- [Background] Johannssen V, Maune S, Werner JA, Rudert H, Ziegler A. Alpha 1-receptors at pre-capillary resistance vessels of the human nasal mucosa. Rhinology. 1997 Dec;35(4):161-5. PMID 9532635
- [Background] Wight RG, Cochrane T. A comparison of the effects of xylometazoline on nasal airflow, and on blood flux as measured by laser Doppler flowmetry. Acta Otolaryngol. 1989 Sep-Oct;108(3-4):284-9. doi: 10.3109/00016488909125529. PMID 2479219
- [Background] Ruffolo RR Jr, Rosing EL, Waddell JE. Receptor interactions of imidazolines. I. Affinity and efficacy for alpha adrenergic receptors in rat aorta. J Pharmacol Exp Ther. 1979 Jun;209(3):429-36. No abstract available. PMID 35606
- [Background] Ruffolo RR Jr, Waddell JE. Receptor interactions of imidazolines: alpha-adrenoceptors of rat and rabbit aortae differentiated by relative potencies, affinities and efficacies of imidazoline agonists. Br J Pharmacol. 1982 Sep;77(1):169-76. doi: 10.1111/j.1476-5381.1982.tb09283.x. PMID 6289955
- [Background] Hein P, Michel MC. Signal transduction and regulation: are all alpha1-adrenergic receptor subtypes created equal? Biochem Pharmacol. 2007 Apr 15;73(8):1097-106. doi: 10.1016/j.bcp.2006.11.001. Epub 2006 Nov 7. PMID 17141737
- [Background] DeBernardis JF, Winn M, Kerkman DJ, Kyncl JJ, Buckner S, Horrom B. A new nasal decongestant, A-57219: a comparison with oxymetazoline. J Pharm Pharmacol. 1987 Sep;39(9):760-3. doi: 10.1111/j.2042-7158.1987.tb06989.x. PMID 2445950
- [Background] Jaillon P. Clinical pharmacokinetics of prazosin. Clin Pharmacokinet. 1980 Jul-Aug;5(4):365-76. doi: 10.2165/00003088-198005040-00004. PMID 6994981
- [Background] Bylund DB, Eikenberg DC, Hieble JP, Langer SZ, Lefkowitz RJ, Minneman KP, Molinoff PB, Ruffolo RR Jr, Trendelenburg U. International Union of Pharmacology nomenclature of adrenoceptors. Pharmacol Rev. 1994 Jun;46(2):121-36. No abstract available. PMID 7938162
- [Background] Hallen H, Enerdal J, Graf P. Fluticasone propionate nasal spray is more effective and has a faster onset of action than placebo in treatment of rhinitis medicamentosa. Clin Exp Allergy. 1997 May;27(5):552-8. PMID 9179430
- [Background] Davies AO, Lefkowitz RJ. Regulation of beta-adrenergic receptors by steroid hormones. Annu Rev Physiol. 1984;46:119-30. doi: 10.1146/annurev.ph.46.030184.001003. No abstract available. PMID 6324653
- [Background] Brodde OE, Brinkmann M, Schemuth R, O'Hara N, Daul A. Terbutaline-induced desensitization of human lymphocyte beta 2-adrenoceptors. Accelerated restoration of beta-adrenoceptor responsiveness by prednisone and ketotifen. J Clin Invest. 1985 Sep;76(3):1096-101. doi: 10.1172/JCI112063. PMID 2995446
- [Background] Tan KS, Grove A, McLean A, Gnosspelius Y, Hall IP, Lipworth BJ. Systemic corticosteriod rapidly reverses bronchodilator subsensitivity induced by formoterol in asthmatic patients. Am J Respir Crit Care Med. 1997 Jul;156(1):28-35. doi: 10.1164/ajrccm.156.1.9610113. PMID 9230722
- [Background] Hamamdzic D, Duzic E, Sherlock JD, Lanier SM. Regulation of alpha 2-adrenergic receptor expression and signaling in pancreatic beta-cells. Am J Physiol. 1995 Jul;269(1 Pt 1):E162-71. doi: 10.1152/ajpendo.1995.269.1.E162. PMID 7631772
- [Background] Hochban W, Althoff H, Ziegler A. Nasal decongestion with imidazoline derivatives: acoustic rhinometry measurements. Eur J Clin Pharmacol. 1999 Mar;55(1):7-12. doi: 10.1007/s002280050585. PMID 10206078
- [Result] Vaidyanathan S, Williamson P, Clearie K, Khan F, Lipworth B. Fluticasone reverses oxymetazoline-induced tachyphylaxis of response and rebound congestion. Am J Respir Crit Care Med. 2010 Jul 1;182(1):19-24. doi: 10.1164/rccm.200911-1701OC. Epub 2010 Mar 4. PMID 20203244
- [Derived] Vaidyanathan S, Williamson P, Lipworth B. Comparative evaluation of nasal blood flow and airflow in the decongestant response to oxymetazoline. Ann Allergy Asthma Immunol. 2012 Feb;108(2):77-80. doi: 10.1016/j.anai.2011.11.013. PMID 22289724